CLINICAL TRIAL: NCT05582031
Title: An Open-label, Phase II, Multi-cohort, 2-stage Trial to Evaluate the Efficacy and Safety of Regorafenib in Combination With Tislelizumab in Patients With Selected Mismatch Repair-Proficient/Microsatellite Stable Pretreated Solid Cancers
Brief Title: Regorafenib With Tislelizumab in Patients With Selected Mismatch Repair-Proficient/Microsatellite Stable Cancers
Acronym: REFIT-MSS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started/ will not proceed.
Sponsor: Translational Research in Oncology (Other)
Collaborators: Bayer (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIO042
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Anal Squamous Cell Carcinoma; Colorectal Neoplasms; Soft Tissue Sarcoma; Malignant Pleural Mesothelioma; Small Cell Lung Carcinoma; Castrate Resistant Prostate Cancer; Neuroendocrine Carcinoma of Prostate; Gastroenteropancreatic Neuroendocrine Neoplasm
Keywords: pMMR; MSS; Advanced solid tumors; MKI; PD-1 inhibitors
MeSH Terms: conditions — Anus Neoplasms; Colorectal Neoplasms; Sarcoma; Mesothelioma, Malignant; Small Cell Lung Carcinoma | interventions — regorafenib; tislelizumab

STUDY DESIGN:
Intervention Model Description: The trial will include 8 cohorts of patients. Each cohort is considered as a single-arm activity-estimating sub-study with PFS-6 as the primary endpoint. A strong primary endpoint signal seen in a cohort may allow for expansion of the cohort, independently of the status of the other cohorts. Similarly, a cohort may be opened and/or closed for enrollment independently of others.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib 90 mg + Tislelizumab 300 mg (Rego-Tisle) (Experimental): The trial will include 8 cohorts of patients, with each cohort considered as a single-arm; all patients enrolled will be treated with regorafenib at a dose of 90 mg orally once daily, on days 1 to 21 of a 28 cycle in combination with tislelizumab 300 mg intravenously day 1 (of a 28 day cycle).
  Interventions: Combination Product: Regorafenib in combination with Tislelizumab

INTERVENTIONS:
Combination Product: Regorafenib in combination with Tislelizumab — Regorafenib 30 mg/tablet + Tislelizumab 100 mg/10 ml vial

SUMMARY:
REFIT-MSS is a non-randomized, multicenter, open-label, multi-cohort, 2-stage, phase II trial to evaluate the efficacy and safety of regorafenib in combination with tislelizumab (referred as Rego-Tisle) in adult patients with select advance, previously treated, Mismatch Repair-Proficient/Microsatellite (pMMR/MSS) stable solid cancers.

The multi-cohort design will allow for the examination of 8 separate cohorts of different cancers to determine whether further examination may be warranted in the individual indications.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, open-label, multi-cohort, phase II trial to evaluate the efficacy and safety of Rego-Tisle in adult patients with solid tumors that are advanced, pretreated and refractory to standard therapy. Approximately 322 evaluable patients (between 15 and 82 per cohort) in around 65 sites will be enrolled to power the trial efficiently to measure the primary endpoint, Progression Free Survival at 6 months (PFS-6).

Patients should have at least one measurable lesion per Response Evaluation Criteria in Solid Tumors guidelines version 1.1 (RECIST 1.1), an Eastern Cooperative Oncology Group Performance Scale (ECOG PS) 0-1, and adequate organ function.

The trial will include patients who had been diagnosed with a histologically or cytologically confirmed solid tumor belonging to any of the types in the cohorts to be enrolled. To be eligible, patient must meet the criteria for tumor type, stage and prior anti-cancer therapy according to inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated PICF obtained prior to any trial-specific procedure that is not part of standard patient care.
2. Patient is ≥ 18 years-old at the time of PICF signature (or the legal age of consent in the jurisdiction in which the trial is taking place).
3. Histologically or cytologically confirmed solid tumor belonging to one of the cohorts specified in the protocol. To be eligible, patient must meet the criteria for tumor type, stage and prior anti-cancer therapy according to the protocol.
4. Tumor must be:

   * In all colorectal (CRC patients) and in any non-CRC patient with dMMR/MSI testing available prior to enrollment: pMMR/MSS tumor based on IHC, MSI-PCR or NGS testing, as performed at the site prior to enrollment according to site's standard practice.
   * In any non-CRC patient with unknown dMMR/MSI status: the site must confirm at screening that the patient has available and retrievable archival tumor tissue from the primary or metastatic site, for submission to a central laboratory for dMMR/MSI testing.
5. Measurable disease by CT or MRI per Response Evaluation Criteria in Solid Tumors (version 1.1), based on tumor assessment performed within 28 days of enrollment.
6. Progressive cancer at the time of trial entry based on clinical or radiographic findings or tumor marker evaluation, according to Investigator's judgment, or cancer that is not amenable to standard therapies even if not progressing.
7. ECOG Performance Scale score of 0 or 1 at enrollment.
8. Adequate hematologic and organ function as assessed by the following laboratory tests, performed at screening (specified within the protocol).
9. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
10. Women of childbearing potential (CBP) must have confirmed negative serum pregnancy test (for β-hCG) within 7 days prior to enrollment.
11. Women of CBP must agree to remain completely abstinent (complete avoidance of heterosexual intercourse) or use highly effective contraceptive methods (i.e., with a failure rate of < 1% per year) during the Treatment Phase and for at least 7 months after the last trial treatment intervention.
12. Men who are sexually active with women of CBP must agree to remain completely abstinent (complete avoidance of heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm during the Treatment Phase and for a total of 7 months post-treatment completion.

Exclusion Criteria:

1. Prior treatment with regorafenib.
2. Prior treatment with a PD1, PD-L1/PD-L2, or CTLA-4 inhibitor, or any other drug or antibody targeting T-cell co-stimulation or checkpoint pathways, except in patients that meet all the following criteria:

   * Patient received a PD1, PD-L1/PD-L2, or CTLA-4 inhibitor, or any other drug or antibody targeting T-cell co-stimulation or checkpoint pathways in either:

     1. Neoadjuvant and/or adjuvant setting and had no relapse within 12 months of completing immunotherapy
     2. Advanced disease setting and had no progression during immunotherapy
   * Patient tolerated immunotherapy and did not need to discontinue treatment due to intolerable toxicity
3. Evidence of progressive or symptomatic CNS metastases. Patients with treated CNS metastases are eligible if they meet all the following criteria:

   * Minimal neurologic symptoms
   * Evidence of stable disease (for at least 2 weeks prior to enrollment) or response on a follow-up scan performed after CNS treatment completion
   * Require corticosteroids at a dose ≤ 10 mg daily of prednisone or equivalent
4. Previous treatment with live vaccine within 28 days of planned start of trial drugs (seasonal flu vaccines that do not contain a live virus are permitted).
5. Concurrent participation in another clinical study, unless it is: (a) an observational (noninterventional) study, or (b) the follow-up period of an interventional trial and patient did not receive an investigational agent/device within 28 days before enrollment (or within 5 half-lives of the drug).
6. Major surgical procedure, open biopsy, significant traumatic injury, radiation therapy and/or systemic anti-cancer therapy ≤28 days prior to enrollment. Patients must have recovered adequately from the toxicity and/or complications from these interventions before enrollment. Radiation therapy given with palliative intent is allowable if finalized ≥ 14 days prior to enrollment.
7. Known hypersensitivity to any of the trial drugs or its formulation components.
8. Active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids.
9. Requirement of systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medications ≤ 14 days prior to enrollment.
10. Uncontrolled diabetes or > Grade 1 laboratory test abnormalities in potassium, sodium, or calcium despite standard medical management or ≥ Grade 3 hypoalbuminemia, ≤ 14 days prior to enrollment.
11. Interstitial lung disease, non-infectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, or clinically significant acute lung diseases.
12. Any cardiovascular conditions as listed within the protocol.
13. Infection requiring systemic (oral or i.v.) antibacterial, antifungal or antiviral therapy ≤14 days prior to enrollment.
14. Patient unable to swallow and retain oral medication or has impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the oral trial treatment (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, small bowel resection).
15. Prior allogeneic stem cell transplantation or organ transplantation.
16. Evidence or history of bleeding diathesis or any hemorrhage or bleeding event > NCI CTCAE v5.0 Grade 3 within 4 weeks prior to enrollment.
17. Non-healing wound, ulcer, or bone fracture.
18. Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 2 years before enrollment. Note: patients with prior or concurrent adequately treated, basal or squamous cell skin carcinoma or adequately treated in situ carcinomas are eligible.
19. Patient has known active HBV or HCV.
20. Patient has HIV infection, unless they meet certain criteria (listed within the protocol).
21. Persistent proteinuria of NCI CTCAE v5.0 Grade 3. Urine dipstick result of ≥ 3+ is allowed if protein excretion (estimated by urine protein/creatinine ratio on a random urine sample) is < 3.5 g/24 hours.
22. Unresolved clinically significant toxicity (per Investigator's assessment) greater than NCI CTCAE v5.0 Grade 1 attributed to any prior therapy/procedure, excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2 (according to NCI CTCAE v5.0).
23. Patient has any other concurrent severe and/or uncontrolled medical condition or personal, psychological, geographic or social circumstance, that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol and retention.
24. Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months (PFS-6) as per Investigator Assessment | 6 Months
  PFS-6 is defined as the proportion of patients who remained free of PFS event (disease progression or death) at 6 months from the date of enrollment.

SECONDARY OUTCOMES:
Overall Response Rate | 24 Months
  Defined as the proportion of patients who have a complete response (CR) or partial response (PR) based on investigator assessment.
Disease Control Rate (DCR) | 24 Months
  Defined as the proportion of patients who have CR, PR, or stable disease (SD) according to RECIST 1.1, as per investigator assessment.
Duration of Response (DOR) | 24 Months
  Defined as the time (in months) from first documentation of response (PR or CR) to progressive disease (PD) or death, based on investigator assessment or death, in patients who had best overall response of CR or PR.
Growth Modulation Index (GMI) | 24 Months
  Defined as as the ratio of time to progression (TTP) with the nth line (TTP(n)) of therapy to the TTP(n)(-1) with the n-1th line.
Overall Survival (OS) | 12 Months
  Defined as time from date of enrollment to date of death due to any cause. Median OS, OS at 6 months (OS-6) and OS at 12 months (OS-12) will be evaluated.
Time to Prostate Specific Antigen (PSA) Progression | 24 Months
  In metastatic castration-resistant prostate cancer (mCRPC) cohort only; defined as the time from the date of enrollment to the date of PSA progression based on Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria
Frequency and Severity of Adverse Events (AEs) and Laboratory Abnormalities | 24 Months
  Frequency and severity of AEs and laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, Study Chair — Medical Oncology Department, Vall d'Hebron Institute of Oncology, CIBERONC